CLINICAL TRIAL: NCT00451646
Title: A Double-blind, Randomised Study Comparing the Safety and Tolerance of SMOFlipid 20% in Long-term Treatment With Parenteral Nutrition
Brief Title: Study Comparing the Safety and Tolerance of SMOFlipid 20% in Long-term Treatment With Parenteral Nutrition
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Dr. Ingrid Mueller, Fresenius Kabi Deutschland GmbH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-SMOF-006
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2008-10

CONDITIONS: Parenteral Nutrition
MeSH Terms: conditions — Hyperphagia | interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): SMOFlipid
  Interventions: Drug: SMOF lipid and Intralipid
- 2 (Active Comparator): Intralipid
  Interventions: Drug: SMOF lipid and Intralipid

INTERVENTIONS:
Drug: SMOF lipid and Intralipid — 1-2 g, 5-7 days, 28 days

SUMMARY:
The aim of this study is to evaluate the safety and tolerance of SMOFlipid 20% in comparison to a standard lipid emulsion Intralipid 20% in patients requiring long-term parenteral nutrition. The safety and tolerance will be evaluated by biochemistry, hematology and coagulation variables, vital signs and adverse events. Further objectives to evaluate are the influence of SMOFlipid 20% on inflammation processes, the efficacy of anti-oxidative properties of vitamin E supplemented to SMOFlipid 20%, and the fatty acid pattern in red blood cells and serum.

ELIGIBILITY:
Inclusion Criteria:

* In- and out-patients in need of parenteral nutrition due to inability to sustain an adequate oral/enteral food intake for at least 4 weeks
* Written consent from the subject

Exclusion Criteria:

* Known hypersensitivity to fish-, egg-, soy-, or peanut-protein or to any of the active substances or excipients
* Known type IV hyperlipidemia, disturbances in lipid metabolism or hypertriglyceridemia
* Severe liver insufficiency
* Severe blood coagulation disorders
* Subjects with chronic stable renal insufficiency defined as S-creatinine value of > 25 mg/l (200 µmol/l) or receiving dialysis/hemofiltration therapy
* General contraindications to infusion therapy: acute pulmonary oedema, hyperhydration
* Unstable conditions
* Unstable angina pectoris
* Acute shock
* Chemotherapy within 4 weeks before start of the trial
* Chemotherapy during the trial
* Subjects for whom the trial treatment is not appropriate
* Female patients must be surgically sterile; or postmenopausal for at least two years; or if of childbearing potential must have a negative serum pregnancy test and must agree to maintain adequate birth control practice during the study.
* Participation in another clinical study with an investigational drug or an investigational medical device within one month prior to start of study or during the study
* Prior inclusion in the present study
* Any other feature that in the opinion of the investigator should preclude study participation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of SMOFlipid 20% assessed by laboratory and clinical parameters (biochemistry, hematology, coagulation), vital signs, adverse events (AEs) as well as inflammation and lipid peroxidation variables | day 0, week 2, week 4

CONTACTS AND LOCATIONS:
Overall Officials: Jon Shaffer, MD, Principal Investigator — Hope Hospital, Manchester, United Kingdom
Locations (12):
- Australia (2):
  - North Shore Private Hospital, Saint Leonards, New South Wales
  - Monash Medical Centre, Melbourne, Victoria
- Denmark (2):
  - Aalborg University Hospital, Department of Medical Gastroenterology, Aalborg
  - Rigshospitalet, Department of Medical Gastroenterology, Copenhagen
- France (2):
  - Hopital Beaujon, Clichy
  - Hopital Edouard Herriot, Unite de Nutrition a Domicile Lyon, Lyon
- Beilinson Medical Center, Department of Surgery "B", Petah Tikva, Israel
- University Medical Center, Nijmegen, Netherlands
- Poland (2):
  - Wydzial Lekarski I Katedra Chirurgii Ogolnej, Krakow
  - Samodzielny Publiczny Szpital Kliniczny im. Prof. W. Orłowskiego, Warsaw
- United Kingdom (2):
  - Hope Hospital, Manchester
  - University Hospital, Queen's Medical Centre, Nottingham